CLINICAL TRIAL: NCT01242384
Title: Prevention of Preterm Birth Using Cervical Pessary in Pregnant Women After Threatened Preterm Labor
Brief Title: Prevention of Preterm Birth Using Cervical Pessary in Pregnant Women After Threatened Preterm Labor(PECEP-RETARD)
Acronym: PECEP-RETARD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maternal-Infantil Vall d´Hebron Hospital (Other)
Responsible Party: Principal Investigator, Maria Goya, MD, PhD, PhD, Maternal-Infantil Vall d´Hebron Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PECEP-RETARD TRIAL
Record Dates: First submitted 2010-09-28; First posted 2010-11-17 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Expectant Management (No Intervention)
- Placement of cervical pessary since 23 weeks until 37 weeks (Experimental)
  Interventions: Device: Device: Silicon ring (Arabin Pessary)

INTERVENTIONS:
Device: Device: Silicon ring (Arabin Pessary) — Placement of a silicon pessary in the vagina, around the cervix.
  Arms: Placement of cervical pessary since 23 weeks until 37 weeks

SUMMARY:
Placement of a vaginal pessary reduces significantly the rate of spontaneous preterm birth in pregnant women with short cervical length after an episode of threatened preterm labour.

ELIGIBILITY:
Inclusion Criteria:

* Minimal age of 18 years
* Episode of threatened preterm labour

Exclusion Criteria:

* Major fetal abnormalities (requiring surgery or leading to infant death or severe handicap)
* Spontaneous rupture of membranes at the time of randomization
* Cervical cerclage in situ
* Active vaginal bleeding
* Placenta previa

Sample size: 336 singleton (168 per arm) and 128 twins (64 per arm).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2008-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Spontaneous delivery before 34 completed weeks | Each 6 months

SECONDARY OUTCOMES:
Birth weight | Each 6 months
Fetal-Neonatal Death | Each 6 months
Neonatal morbidity | Each 6 months
Maternal adverse effects | Each 6 months
Preterm birth before 37 weeks or 28 weeks | Each 6 months
Rupture of membranes before 34 weeks | Each 6 months
Hospitalisation for threatened preterm labour | Each 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elena Carreras, Study Director — Hospital Vall d'Hebron; Maria Goya, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Vall d'Herbron, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Abdel-Aleem H, Shaaban OM, Abdel-Aleem MA, Aboelfadle Mohamed A. Cervical pessary for preventing preterm birth in singleton pregnancies. Cochrane Database Syst Rev. 2022 Dec 1;12(12):CD014508. doi: 10.1002/14651858.CD014508. PMID 36453699
- [Derived] Merced C, Goya M, Pratcorona L, Rodo C, Llurba E, Higueras T, Cabero L, Carreras E; PECEP-RETARD Trial Group. Cervical pessary for preventing preterm birth in twin pregnancies with maternal short cervix after an episode of threatened preterm labor: randomised controlled trial. Am J Obstet Gynecol. 2019 Jul;221(1):55.e1-55.e14. doi: 10.1016/j.ajog.2019.02.035. Epub 2019 Feb 28. PMID 30826339